CLINICAL TRIAL: NCT01029990
Title: Randomized Controlled Trial to Study Interventions to Increase Participation in Cervical Cancer Screening Program
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Assar Gabrielsson Cancer Foundation, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: OCGbgSw0101
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: participation; mass screening; cervical neoplasia; health economics; cost-benefit
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telephone arm (Experimental): A midwife tries to contact the woman by telephone and offer her an appointment for a PAP-smear
  Interventions: Other: Telephone arm
- Self-test arm (Experimental)
  Interventions: Other: Self-test arm
- Control arm (No Intervention): No intervention other than what is routine in the screening program

INTERVENTIONS:
Other: Telephone arm — Midwifes at 72 antenatal care units in West region of Sweden receive lists with names and telephone numbers on women who have no record of screening during two screening rounds (6 - 10 years depending on age). The midwife will make up to ten attempts to reach each woman and is instructed to use no more than 30 minutes on this. If the midwife get in touch with the woman she will encourage participation in regular screening (run by midwives in Sweden) and help the woman to get an appointment.
  Arms: Telephone arm
Other: Self-test arm — Women receive an offer to order a vaginal self test for HPV. The woman can return a coupon in a postage free envelope and she will receive a self testing kit (dry method) within a couple of days. She will return the test in another postage free envelope. A reminder will be sent to women who order a test but do not return it.
  Arms: Self-test arm

SUMMARY:
Women who don't participate in Swedish cytology screening program are a minority of about 10%, but constitute the majority of those who acquire cervical cancer. Over 50 000 women in the Västra Götalandregion have abstained from participation in the program for at least 2 screening rounds (6 - 10 years, depending om age). We plan to test two promising strategies to increase participation. In a study of two different health policies women who have defaulted are randomised to receiving a telephone call from a midwife, receive an offer of a self-test for HPV or being included in a control group. This is an effectiveness study that should give an answer how participation could be increased and give the basis for a calculation of the costs involved, before decisions can be made about implementing either intervention.

DETAILED DESCRIPTION:
Background

Cervical cancer today is considered as a disease that to a very large extent is preventable. In Sweden cytological screening has been ongoing since the 60:s and this has made cervical cancer a rare disease. Several new, but costly, methods like HPV-testing and vaccination has been claimed to further reduce cancer incidence, but this has not been scientifically proven so far. A recent audit of the Swedish screening program (Andrae 2008) found that the foremost risk factor for cervical cancer in the context of the program was non participation. Women who do participate are well protected from cervical cancer.

A Swedish study evaluating different strategies to increase participation found telephone contact with defaulters to be the superior intervention (Eaker 2004). This study was done in a region of Sweden with lower coverage (Sparén 2007) and less emphasis on efforts to increase participation. A study from Kalmar, Sweden, with high coverage did not find an extended yield to requests from non-participating women to be cost effective (Oscarsson 2007). Self testing for HPV has been advocated as an effective method and there is a kit commercially available (Stenvall 2007). The procedure is used as a routine in Uppsala county and marketed to other counties.

Aim To study two possible interventions to increase participation

Design Randomised controlled trials of two interventions and a control arm

Hypothesis

Intervention with a) supportive telephone contact, by a midwife, with women who do not have a smear registered for two screening rounds will increase participation, increase uptake of precancerous lesions (CIN2+) and is cost effective. b) selftesting for oncogenic papillomavirus (HPV) will increase participation and is cost effective.

Method: selection of study base

Selection was done by random among women aged 29 - 63 who did not have a pap-smear registered within the two recent screening rounds. Women who were excluded from invitation due to total hysterectomy and women who could be identified as have immigrated into the region under the period were excluded before randomisation. July 1 2008 there was 52362 women who fulfilled the first criteria (before exclusions) identified through the Register for Prevention of Cervical Cancer in West Sweden. 8800 selected women will be included and randomised to one of three arms with the distribution 5:1:5

Methods: Intervention Arm A: 4000 randomised women fulfilling inclusion criteria receive a letter informing them they will be contacted by a midwife by phone, to be offered an appointment to take a smear. They can at that stage decline such contact or if they wish return contact information (telephone number). A week later the women who have not declined will be called by a midwife and offered an appointment for taking a smear. Abnormal smear will be followed up with referral to a gynecologist in concordance with normal screening routine.

Arm B: 800 women will be sent an offer of HPV-self sampling (Aprovix, Uppsala, Sweden). By regular mail the woman can order a test kit, and return this to the laboratory after sampling. The samples will be tested with Hybrid Capture II for high risk HPV. A negative result will be communicated to the women. A positive result will be sent to the gynecological clinic responsible for the work up of abnormal cytological screening smears in the area were the woman lives. The afflicted woman will get information from the clinic and an appointment for colposcopy and cytology. Further investigation will be conducted as clinical routine. Reminders will be sent to women who have ordered the kit and not returned any sample. In order to evaluate the effect of a primary reminder women who have not responded to the primary offer within 60 days will receive a reminder.

Arm C (controls) 4000 women will be controls. No specific action will be taken within the study outside routine in the screening program (yearly written reminder when smears are not found in the database)

Methods: Data collection All data about cytology, colposcopy with biopsies and treatment for CIN are registered as a routine in the West Sweden Registry for Cervical Cancer Prevention and data will be extracted from that registry. Data about HPV-testing will be transferred to this registry from the Aprovix laboratory in Uppsala. Man-time needed and costs for material and analyses for the different interventions will be registered as base for health economic assessments.

Primary outcomes: Frequency of testing (cytology in arm A and C and HPV-test in arm B). Frequency of further assessment of abnormal tests (all arms).

Secondary outcomes: (Arm A vs arm C) Frequency of abnormal smears. Frequency of treated CIN, (CIN1, CIN2 and CIN3, grouped as low grade (CIN1) and high grade (CIN2, CIN3, AIS and invasive cancer). Number of invasive cancers and FIGO stadium. Cost of interventions. Cost per CIN2+ found. The study is powered to find a 30% difference in primary outcome based on an expected 20% participation rate in the control group with 80% power at a significance level of 5% for both interventions (A and B compared with C). An expected rate of abnormal smears of 7% among these women with no smear recorded 6 or more years will give a 80% power to find a 60% relative difference in number of abnormal smears (RR=1,6) when intervention arm A is compared with the controls in arm C.

The results from work up of abnormal tests in arm A will be considered representative for arm B as well, given the same level of abnormality.

The cost per participant and per biopsy with CIN found will be calculated. The cost per found and treated high grade CIN will be compared with a reference of estimated €3500 (preliminary figure) per CIN2+ that is eradicated.

Methods:Statistical analysis All analysis will be based on intention to treat. Pearson's Chi2 and Fischers exact test will be used to compare distribution of categorical variables between the groups. One way variances will be used to test differences of means between groups for continuous variables. The cumulated probability for outcome vs. follow up time will be calculated with Kaplan-Meier analysis. Multiple Cox regression will be used to determine relative risks. 95 % confidence intervals will be used throughout and level of significance will be calculated two sided as 5%

ELIGIBILITY:
Inclusion Criteria:

* No record of PAP smear in the regional screening register for more than two screening rounds (6 - 10 years depending on age).
* Evidence in the regional population register that women have been living in the west region of Sweden during this time.

Exclusion Criteria:

* Total hysterectomy

Ages: 29 Years to 63 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8800 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Frequency of testing (cytology in arm A and C and HPV-test in arm B). F | 7 months after invitation
Frequency of further assessment of abnormal tests | 7 months

SECONDARY OUTCOMES:
Frequency of abnormal smears. (Arm A vs arm C) | 7 months
Frequency of treated CIN (Arm A vs. arm C) | 7 months
Number of invasive cancers detected classified by FIGO stadium. | 7 months
Cost of interventions | 7 months
Cost per CIN2+ found and treated | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Björn Strander, MD, PhD, Principal Investigator — Göteborg University